CLINICAL TRIAL: NCT05802316
Title: Awake Tracheal Intubation is Associated With Fewer Adverse Events in Critical Care Patients Than Standard Tracheal Intubation
Brief Title: Awake Tracheal Intubation in Critical Care Patients
Acronym: Awake
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUK
Record Dates: First submitted 2023-03-22; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Videolaryngoscopy; Intensive Care Unit Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- awake: awake tracheal intubation
  Interventions: Device: tracheal intubation using videolaryngoscope with a hyperangulated blade or standard intubation videolaryngoscopy (VL) and direct laryngoscopy (DL)
- asleep: standard intubation videolaryngoscopy (VL) and direct laryngoscopy (DL)
  Interventions: Device: tracheal intubation using videolaryngoscope with a hyperangulated blade or standard intubation videolaryngoscopy (VL) and direct laryngoscopy (DL)

INTERVENTIONS:
Device: tracheal intubation using videolaryngoscope with a hyperangulated blade or standard intubation videolaryngoscopy (VL) and direct laryngoscopy (DL) — In the awake group tracheal intubation performed by an videolaryngoscope with a hyperangulated blade. In the asleep group the standard intubation were performed by videolaryngoscopy (VL) and direct laryngoscopy (DL)

SUMMARY:
Tracheal intubation in critical care is a high-risk procedure requiring significant expertise and airway strategy modifications, such as awake intubation with video laryngoscope or flexible endoscope intubation. Furthermore, delayed sequence intubation can be used by experts in certain high-risk subgroups. The investigators hypothesise that awake tracheal intubation is associated with a lower incidence of severe adverse events than standard tracheal intubation in critical care patients.

DETAILED DESCRIPTION:
Intubation records from 2020 to 2022 were acquired to examine all tracheal intubations of critical care patients at a tertiary hospital. Each awake tracheal intubation (awake) case - all of which were performed using a videolaryngoscope with a hyperangulated blade - was propensity matched with two controls (1:2 ratio; standard intubation videolaryngoscopy (VL) and direct laryngoscopy (DL) undergoing general anaesthesia), with similar comorbidities and intubations performed after the induction of anaesthesia (asleep).

ELIGIBILITY:
Inclusion Criteria:

* Data for all critical care patients requiring tracheal intubation during the study period

Exclusion Criteria:

* included incomplete data reports

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: critical care patients requiring tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Hypotension | during intubation procedure (within 30 Minutes)
  defined as a mean arterial pressure < 55 mmHg
cardiac arrest | during intubation procedure (within 30 Minutes)
  defined as a peri-interventional cardiac arrest
desaturation | during intubation procedure (within 30 Minutes)
  defined as SpO2 < 80% after sufficient preoxygenation

SECONDARY OUTCOMES:
Cormack and Lehane classification (Class I-IV) | during intubation procedure (< 120 seconds)
  glottis visualisation
FPS | during intubation procedure (< 120 seconds)
  First Pass Intubation success
Airway Injury | during intubation procedure (< 120 seconds)
  dental injury
other adverse events | during intubation procedure (< 120 seconds)
  soft tissue injury

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, Principal Investigator — University Medical Centre Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany